CLINICAL TRIAL: NCT05675761
Title: A Prospective, Multicenter, Real World Study to Evaluate the Efficacy and Safety of Azovudine in the Treatment of COVID-19
Brief Title: The Efficacy and Safety of Azovudine in the Treatment of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Innovation-A
Record Dates: First submitted 2023-01-04; First posted 2023-01-09 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Infections; Morality; Death, Assisted
MeSH Terms: conditions — COVID-19; Infections; Suicide, Assisted | interventions — azo rubin S

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Combined bacterial and fungal infection: Combined bacterial and fungal infection
  Interventions: Drug: Azorubine
- No bacterial and fungal infection: No bacterial and fungal infection
  Interventions: Drug: Azorubine

INTERVENTIONS:
Drug: Azorubine — Azovudine tablets, 1mg /tablet, 5 tablets, QD+basic treatment (14 days at most)
  Other Names: basic treatment

SUMMARY:
This study is a prospective, multicenter clinical study. It is intended to discuss the efficacy of starting Azovudine treatment as early as possible for all types of patients of COVID-19, the time of remission of specific symptoms, the proportion of patients with severe diseases, oxygen and conditions, and related adverse reactions, so as to understand the efficacy and safety of Azovudine treatment in all types of COVID-19, and provide real world data support for the treatment of the majority of COVID-19 patients.

DETAILED DESCRIPTION:
1. To evaluate the clinical efficacy of Azovudine in the treatment of mild, moderate and severe COVID-19.
2. To explore the safety and adverse reactions of Azovudine in the whole population of COVID-19.
3. To explore the remission time of clinical symptoms, signs and images of patients with COVID-19 treated with Azovudine.
4. Explore the clinical guiding value of CORMB score.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old;
2. Respiratory tract samples (nasopharynx, oropharynx, lower respiratory tract [such as sputum]) collected within 96 hours before enrollment were confirmed to be SARS CoV-2 positive by RT-PCR virus molecular amplification;
3. At least one symptom or sign of COVID-19 (symptoms and signs related to COVID-19, including cough, expectoration, dyspnea, fever, chills, fatigue, muscle soreness, diarrhea, headache, sore throat, nasal congestion, runny nose, etc.);
4. Participants who meet one or more of the following requirements: from the first COVID-19 symptom to the first medication ≤ 5 days;
5. Agree to observe contraceptive measures during the clinical trial;
6. Participants who understand and agree to follow the planned research procedures;
7. Provide follow-up information during the study;
8. Understand the study and be willing to sign the informed consent form.

Exclusion Criteria:

1. Those who are known to be allergic to any component of the intervention preparation used in the test;
2. Patients with abnormal liver function test (alanine aminotransferase and /or glutamic oxaloacetic aminotransferase exceed the upper limit of normal value by 3 times, or total bilirubin exceeds the upper limit of normal value by 2 times);
3. Patients with a known history of liver disease (cirrhosis with ChildPugh grade B and C);
4. Congestive heart failure within 6 months (NYHA ¾ Grade), patients with untreated symptomatic arrhythmia or myocardial infarction history;
5. Individuals with malabsorption syndrome or other diseases affecting gastrointestinal absorption, and patients who need intravenous nutrition or cannot take orally or through nasogastric tube;
6. Participants who have received other SARS CoV-2 monoclonal antibody therapy or antiviral therapy (including research therapy);
7. Participants who received COVID-19 convalescent plasma therapy;
8. Patients receiving anti HIV treatment;
9. Participants who also participate in any other type of medical research or are considered to be scientifically or medically incompatible with this research;
10. Participants who have participated in the intervention clinical research in the past 30 days should pass 5 half lives or 30 days, whichever is longer, if the previous research intervention has a longer half life.
11. Researchers believe that the test will endanger any health and safety of participants;
12. Women who are pregnant, nursing or planning to be pregnant during the study period or men whose partners plan to be pregnant during the study period;
13. Unable to provide informed consent.Contacts and Locations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with novel coronavirus infection meeting the criteria of The New Coronavirus Pneumonia Diagnosis and Treatment Program (Ninth Edition)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Continuous recovery time of clinical symptoms of Azovudine in the treatment of COVID-19 | Day 1 to 28 days
  Continuous recovery time of clinical symptoms of Azovudine in the treatment of COVID-19
Safety evaluation results: for example, AE (adverse events) and SAE (serious adverse events) up to the 28th day | Up to 28 days
  Safety evaluation results: for example, AE (adverse events) and SAE (serious adverse events) up to the 28th dayof Novel Coronavirus Infection by the National Health Commission (Trial Version 9) The development from asymptomatic to mild/general-type The development from mild to general-type/severe type The development from general-type to severe/critical type The development from severe to critical type

SECONDARY OUTCOMES:
Evaluation of positive rate | Day 1 to 28 days
  nucleic acid and /or antigen retest is positive within 28 days after negative conversion of nucleic acid and /or antigen

CONTACTS AND LOCATIONS:
Overall Officials: zongyang yu, Ph.D, Principal Investigator — The 900th Hospital of the Joint Logistic Support Force, PLA
Locations (1):
- The 900th Hospital of the Joint Logistic Support Force, PLA, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No